CLINICAL TRIAL: NCT00597077
Title: Atrial Fibrillation and Congestive Heart Failure (AF-CHF)Trial
Brief Title: Atrial Fibrillation and Congestive Heart Failure Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Denis Roy, MD, Montreal Heart Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 41552; ISRCTN84858671
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Last update posted 2008-02-08 (Estimated); Status verified 2008-01

CONDITIONS: Atrial Fibrillation; Congestive Heart Failure
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rate control (Active Comparator)
  Interventions: Other: Rate vs rhythm control strategies for atrial fibrillation
- Rhythm control (Active Comparator)
  Interventions: Other: Rate vs rhythm control strategies in atrial fibrillation

INTERVENTIONS:
Other: Rate vs rhythm control strategies for atrial fibrillation — Rate vs rhythm control strategies for atrial fibrillation
  Arms: Rate control
Other: Rate vs rhythm control strategies in atrial fibrillation — rate vs rhythm control strategies in atrial fibrillation
  Arms: Rhythm control

SUMMARY:
Heart failure is a clinical syndrome where the heart is unable to pump enough blood to satisfy the organism's metabolic needs. Heart failure has become a major clinical and public health problem with approximately 300,000 Canadians being affected. Atrial fibrillation is a rhythm disorder in which the upper chambers of the heart (the atria) are paralyzed by continuous electrical activity. Some of the continuous chaotic electrical activity in the atria travels to the lower cavities of the heart (the ventricles) causing then to beat irregularly and very rapidly. It is the most frequent cardiac arrhythmia, affecting 5% of individuals 65 years and older and it is associated with an increased risk of stroke. Both conditions (heart failure and atrial fibrillation) often co-exist in the same patient. Heart failure promotes atrial fibrillation and atrial fibrillation aggravates heart failure. The Atrial Fibrillation and Congestive Heart Failure (AF-CHF) trial is investigating whether preservation of normal cardiac rhythm influences mortality and morbidity. The AF-CHF study began in 2001 and 1,378 patients have been enrolled from 123 participating centres, in North America, South America, Europe, and Israel. The results of this trial which are expected in October 2007, will improve decision-making for the physician and will provide useful information to healthcare organizations responsible for the care of heart failure patients.

DETAILED DESCRIPTION:
Congestive heart failure (CHF) and atrial fibrillation (AF) are two important and growing problems in medicine and cardiology. Both conditions often co-exist and complicate each other's management. Two therapeutic strategies are available for patients with AF and CHF: the first aims at restoring and maintaining sinus rhythm, whereas, the second focuses exclusively on optimizing ventricular rate. The primary objective of the Atrial Fibrillation and Congestive Heart Failure (AF-CHF) trial is to compare these two widely-used treatment strategies with respect to cardiovascular mortality.

Hypothesis: Restoring and maintaining sinus rhythm reduces cardiovascular mortality compared to a rate control treatment strategy in patients with AF and CHF.

Rationale: Despite new therapeutic interventions, the prognosis of heart failure patients remains grim with 5-year survival rates usually less than 50%. In most recent, large CHF trials, AF has been reported to be independently associated with increased mortality. Non-randomized observations also suggest that patients with AF in the setting of CHF have a greater tendency to revert to sinus rhythm during amiodarone therapy or with newer class III antiarrhythmic agents and that those who maintain a normal rhythm have a better prognosis. There is a need to determine whether a treatment strategy that attempts to maintain sinus rhythm will have a beneficial impact on cardiovascular mortality in CHF patients. This hypothesis has never been tested in a prospective, controlled, adequately-powered randomized trial.

Research Plan: AF-CHF is a prospective, multicentre clinical trial (100 centres in Canada, the USA, and Europe), that will randomize 1,450 NYHA class II-IV CHF patients with left ventricular ejection fraction >/=35% (NYHA class I patients with prior hospitalization for CHF or ejection fraction </=25% are also eligible) and a history of significant AF (ECG documentation of either one episode lasting >/=6 hours within the past 6 months, or an episode lasting >/=10 minutes within the past 6 months in a patient with prior electrical cardioversion for AF) to one of two treatment strategies: 1) rhythm control with the use of electrical cardioversion if needed combined with antiarrhythmic drug therapy (amiodarone or other class III agents), and additional non-pharmacologic therapy in resistant patients, 2) rate control with the use of drugs (mainly beta-blockers plus digoxin) and/or pacemaker and AV nodal catheter ablation if necessary. The enrollment period will be completed within 2 years with a minimum follow-up of 2 years. Both groups will receive optimal CHF management with ACE inhibitors and beta-blockers. Cardiovascular mortality will be the primary endpoint of the trial. The intention-to-treat approach will be the primary method of analysis. Secondary outcomes are total mortality, hospitalization, stroke, cost of therapy and quality of life. From recent trial data, we anticipate a 18.75% 2-year cardiovascular mortality in the rate control arm and a 25% reduction in cardiovascular mortality in the rhythm control group. Assuming a 2% loss to follow-up, a two-sided alpha level of 0.05 and an annual accrual rate of 750 patients, we calculate that 722 patients per group (rounded total number of 1,450 patients) will be necessary to achieve a power of 0.80 when performing a log-rank test. The Research Centre of the Montreal Heart Institute will be the Coordinating and Methods Centre.

ELIGIBILITY:
Inclusion Criteria:

1. Left ventricular ejection fraction </=35% as measured by nuclear imaging, echocardiography, or cardiac angiography within 6 months preceding enrollment. If the patient has had a myocardial infarction or heart surgery during this period, the ejection fraction must be remeasured.
2. Symptomatic CHF (NYHA class II-IV) at some time during the 6 months before randomization, despite therapy with an ACE inhibitor (however, patients who do not tolerate an ACE inhibitor are eligible). Asymptomatic patients (NYHA class I) with either a prior hospitalization for CHF during the 6 months before randomization or with a left ventricular ejection fraction of </=25% are also eligible.
3. History of significant AF, defined as either:

   1. one episode lasting >/=6 hours (duration of AF will be determined by history), within the past 6 months with electrocardiographic confirmation; or
   2. an episode lasting >/=10 minutes (by history) within the past 6 months with electrocardiographic confirmation in a patient with a prior electrical cardioversion for AF.
4. In the opinion of the clinical investigator, the patient must be eligible for long-term treatment with either treatment strategy of AF.

Exclusion Criteria:

1. AF is known to be present and uninterrupted for more than 12 months prior to randomization. However, if such a patient is cardioverted and maintained in sinus rhythm for >/=24 hours, he or she becomes eligible.
2. Reversible cause of AF such as acute pericarditis, pulmonary embolism, hyperthyroidism, alcohol intoxication.
3. AF occurring and not persisting beyond 10 days of surgery or myocardial infarction.
4. Reversible cause of CHF such as severe aortic or mitral stenosis and tachycardia-induced cardiomyopathy.
5. Decompensated CHF within 48 hours of randomization.
6. Antiarrhythmic drugs other than calcium channel blockers, beta-blockers or digoxin required for other arrhythmias or other indications.
7. More than 7 days of amiodarone therapy within the last month prior to randomization.
8. Second or third degree AV block, sinus pause >3 seconds, resting heart rate <50 bpm without a permanent pacemaker.
9. History of drug-induced Torsades de Pointes or congenital long QT syndrome.
10. Prior AV nodal ablation or Maze surgery.
11. Probable cardiac transplantation in the next 6 months.
12. Chronic renal failure requiring dialysis.
13. Women of child-bearing potential and not on a reliable method of birth control.
14. Geographic or social factors, drug or alcohol abuse making follow-up or compliance difficult.
15. Other noncardiovascular medical condition (such as cancer) making 1 year survival unlikely.
16. Less than 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1376 (Actual)
Dates: Start 2001-04; Primary Completion 2007-06 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
cardiovascular death | Minimum of 2 years and a maximum of 6 years

SECONDARY OUTCOMES:
Total mortality | Minimun of 2 years and a maxiumum of 6 years
Stroke | Minimum of 2 years and a maximum of 6 years
Worsening CHF | Minimum of 2 years and maximum of 6 years
Hospitalization | Minumum of 2 years and maximum of 6 years
Composite endpoint of CV death and worsening CHF | Minimum of 2 years and a maximum of 6 years
Composite endpoint of CV death, stroke and worsening CHF | Minimum of 2 years and a maximum of 6 years
Quality of life/depression | Minimum of 2 years and a maximum of 6 years
Cost of therapy | Minimum of 2 years and a maximum of 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Denis Roy, Study Director — Montreal Heart Institute
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

REFERENCES:
- [Derived] O'Meara E, Khairy P, Blanchet MC, de Denus S, Pedersen OD, Levesque S, Talajic M, Ducharme A, White M, Racine N, Rouleau JL, Tardif JC, Roy D; AF-CHF investigators. Mineralocorticoid receptor antagonists and cardiovascular mortality in patients with atrial fibrillation and left ventricular dysfunction: insights from the Atrial Fibrillation and Congestive Heart Failure Trial. Circ Heart Fail. 2012 Sep 1;5(5):586-93. doi: 10.1161/CIRCHEARTFAILURE.111.965160. Epub 2012 Jul 12. PMID 22798522
- [Derived] Frasure-Smith N, Lesperance F, Habra M, Talajic M, Khairy P, Dorian P, Roy D; Atrial Fibrillation and Congestive Heart Failure Investigators. Elevated depression symptoms predict long-term cardiovascular mortality in patients with atrial fibrillation and heart failure. Circulation. 2009 Jul 14;120(2):134-40, 3p following 140. doi: 10.1161/CIRCULATIONAHA.109.851675. Epub 2009 Jun 29. PMID 19564557
- [Derived] Roy D, Talajic M, Nattel S, Wyse DG, Dorian P, Lee KL, Bourassa MG, Arnold JM, Buxton AE, Camm AJ, Connolly SJ, Dubuc M, Ducharme A, Guerra PG, Hohnloser SH, Lambert J, Le Heuzey JY, O'Hara G, Pedersen OD, Rouleau JL, Singh BN, Stevenson LW, Stevenson WG, Thibault B, Waldo AL; Atrial Fibrillation and Congestive Heart Failure Investigators. Rhythm control versus rate control for atrial fibrillation and heart failure. N Engl J Med. 2008 Jun 19;358(25):2667-77. doi: 10.1056/NEJMoa0708789. PMID 18565859